CLINICAL TRIAL: NCT03807518
Title: The Effect of a Pre- and Post- Operative Exercise Programme Versus Standard Care on Physical Fitness in People With Upper Gastrointestinal Cancers- Study Protocol for a Randomised Control Trial: The PERIOP-OG Trial.
Brief Title: Pre- and Post-Operative Exercise Program in Upper Gastrointestinal Cancers
Acronym: PERIOP-OG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal College of Surgeons, Ireland (Other)
Collaborators: Beaumont Hospital (Other); Mercy University Hospital, Cork, Ireland (Other); Dublin City University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: RCSI 18/58
Record Dates: First submitted 2018-12-17; First posted 2019-01-17 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2020-05

CONDITIONS: Exercise Intervention
Keywords: Oesophageal Cancer; Gastric Cancer; Physical Fitness
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms

STUDY DESIGN:
Intervention Model Description: Parallel group randomised 1:1 controlled multi centre trial
Who Masked: Investigator
Masking Description: The investigator will be blinded to the allocation of the participants
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Structured Exercise Intervention (Experimental): The exercise training program was designed to improve physical fitness while the patients are receiving neoadjuvant treatment prior to surgery and for a 6 week period after surgery once patients are deemed fit to return to training.
  Interventions: Behavioral: Standard Exercise Program
- Standard Oncological Care (No Intervention): This group will receive standard oncological care and will receive no formal education of exercise intervention.

INTERVENTIONS:
Behavioral: Standard Exercise Program — Standard Exercise Program- Participants will be invited to take part in a structured home, supervised, or both, exercise program while undergoing neo adjuvant therapy and for a six week period when deemed fit post surgery.
  Arms: Structured Exercise Intervention

SUMMARY:
Esophageal and gastric cancers are a considerable health burden. In the past 10 years the 5-year survival for both cancers has doubled. This is due to a number of factors including advances in neo adjuvant and adjuvant chemotherapy and radiotherapy. However, physical fitness significantly declines as a result of neo adjuvant an adjuvant therapy. From studies in other cancers it is known that peri operative training improves physical fitness, yet there is little research into its effects in those with upper gastrointestinal cancers. The aim of this study is to assess the effect of a pre-and post operative training program on patients with upper gastrointestinal cancers on their physical fitness and consequently their optimism, quality of life and post operative morbidity.

DETAILED DESCRIPTION:
The comparator in this study will be standard oncological care. There patients will receive the exact same care as the intervention group patients but will receive no exercise training program.

The primary goal of this multi-centre randomised controlled trial are to investigate the effects of peri-operative exercise training programmes on physical fitness, measured with a 6 minute walk test, in patients undergoing a major curative upper-GI resection for either oesophageal or gastric cancer.

The secondary aims will look at the effect of peri-operative exercise training on patients quality of life, optimism and well being, post operative morbidity, nutritional status and blood markers of inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years of age or above;
* Have confirmed Multi Disciplinary Team (MDT) evidence of adenocarcinoma or squamous cell cancer of the oesophagus, oesophago- gastric junction or stomach requiring neoadjuvant therapy and planned curative resection.
* Be referred by a multidisciplinary team meeting for neo adjuvant chemotherapy or neo adjuvant chemoradiotherapy prior to planned oesophagectomy or gastrectomy.
* Have measurement confirming (endoscopic or otherwise) that the tumour starts more than 5cm below cricopharyngeus;
* Be fit for pre-operative anaesthesia and surgery
* Be able to provide written informed consent.

Exclusion Criteria:

* Inability to participate in the exercise program (unable to perform 6 Minute Walk Test, unable to attend for assessment of parameters at any time point).
* Patients with high grade dysplasia (squamous cell or adenocarcinoma);
* Patients who have or develop metastatic disease at time of enrolment or during their neoadjuvant therapy;
* Patients being referred for primary surgery without requirement for neoadjuvant treatment;
* Patients with squamous cell cancer of the oesophagus who the MDT recommends or who individually elect to undergo definitive chemoradiotherapy;
* Evidence of previous/concomitant malignancy that would interfere with this treatment protocol;
* Pregnancy;
* Patients participating in other trials that would interfere with the implementation of this protocol at a particular site.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-12-19 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Change in Physical Fitness | Baseline, one week after completion of neo adjuvant treatment, one week before surgery, six weeks after surgery, twelve weeks after surgery
  The primary goal of this multi-centre randomised controlled trial is to investigate the effects of peri-operative exercise training programmes on physical fitness, defined as the distance covered in metres and centimetres during a 6 minute walk test, in patients undergoing a major curative upper-GI resection for either oesophageal or gastric cancer. To complete the Six Minute Walk Test, no warm up is permitted and participants rest in a seated position for 10 minutes prior to the test beginning. Participants walk up and down a 20m course marked by cones for 6 minutes under instruction to cover as much ground as possible. The number of laps completed is recorded. A standard set of instructions as well as encouragement is used. After 6 minutes, the participant stops and the distance covered in the final partial lap as measured and total distance covered is calculated. Change from baseline to post treatment difference between groups.

SECONDARY OUTCOMES:
Change in Strength - The Sit to Stand Test | Baseline, one week after completion of neo adjuvant treatment, one week before surgery, six weeks after surgery, twelve weeks after surgery
  Strength will be measured using two tests. the Sit to Stand Test . Participants will sit on a chair (height 43-45 cm) with arms crossed on their, and legs flat on the floor, parallel to each other, and approximately shoulder width apart. Participants will stand up and sit down 10 times as quickly as possible. Participants must not bounce off the chair when moving from a seated position to standing position. They must fully extend their legs on each stand. The time taken to perform 10 repetitions will be timed using a stopwatch. Participants will perform two trials and the best trial will be recorded as their score. Change from baseline to post treatment difference between groups.
Change in Strength - The Handgrip Test | Baseline, one week after completion of neo adjuvant treatment, one week before surgery, six weeks after surgery, twelve weeks after surgery
  Strength will be measured using a hand dynamometer. The test will be conducted in a standing position with the upper arm tight against the participant's trunk and the forearm at a right angle to the upper arm. If this is not possible the participant may sit in an upright chair or use their free hand to rest the dynamometer on a table to support the arm. The gripping handle will be set to a comfortable width to ensure the patient can rest the middle piece of the fourfingers on the handle. The participant will be instructed to squeeze the handle with maximum force for a few seconds. The value on the scale will be recorded. The participant will complete two trials on each hand. The highest score will be accepted.Change from baseline to post treatment difference between groups.
Change in Body Composition | Baseline, one week after completion of neo adjuvant treatment, one week before surgery, six weeks after surgery, twelve weeks after surgery
  Determined by body mass index (BMI). BMI will be calculated as weight in kilograms divided by height in meters squared. Height will be measured using a wall stadiometer to the nearest .1cm. Weight will be measured using an electronic scales to the nearest .1kg.Change from baseline to post treatment difference between groups.
Change in Physical Activity - Accelerometer | Baseline, one week after completion of neo adjuvant treatment, one week before surgery, six weeks after surgery, twelve weeks after surgery
  This will be measured using two assessments: 3-day ActivPAL3 triaxial accelerometer. Participants will be instructed to wear the device on the midpoint of the anterior aspect of the right thigh and attach using a film adhesive frame dressing. They will continue to wear this for three days continuously. They cannot wear the ActivPAL3 triaxial accelerometer during water activity periods. Change from baseline to post treatment difference between groups.
Change in Quality of Life measured using the EQ-5D Health Questionnaire | Baseline, one week after completion of neo adjuvant treatment, one week before surgery, six weeks after surgery, twelve weeks after surgery
  EQ-5D (Euro qual health questionnaire consists of 5 themes graded 1-5 and an overall score. The questionnaire is then converted to an index value using the Crosswalk value sets developed for the EQ-5D Health Questionnaire.
  There is a descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, extreme problems. The respondent is asked to indicate his/her health state by ticking (or placing a cross) in the box against the most appropriate statement in each of the 5 dimensions.
  The EQ VAS records the respondent's self-rated health on a 20 cm vertical, visual analogue scale with endpoints labeled 'the best health you can imagine' and 'the worst health you can imagine.
Change in Optimism | Baseline, Change from baseline to one week before surgery
  Optimism as an outcome is measured using the Life Orientation Test-Revised (LOT-R: Scheier, Carver, & Bridges, 1994) and consists of ten items assessing generalised expectancies for positive versus negative outcomes. This will be administered at baseline and pre-surgery only. The scale uses 10 questions on a 1-10. There are 4 filler questions. High scores indicate optimism.
Change in Well Being-The Functional Assessment of Cancer Therapy (FACT-E) questionnaire. | Baseline, one week after completion of neo adjuvant treatment, one week before surgery, six weeks after surgery, twelve weeks after surgery
  Functional Assessment of Cancer Therapy-Esophageal (FACT-E) questionnaire. This is an HRQOL instrument validated in patients with esophageal cancer. It is composed of a general component (FACT-G) and an esophageal cancer subscale (ECS). Patients will score a series of questions (0 = not at all; 4 = very much) in five sections (physical well-being; social/family well-being; emotional well-being; functional well-being; additional concerns) for the past 7 days. Higher scores will suggest better quality of life.
Well Being - Semi-structured Interviews. | One week before surgery
  Semi-structured interviews will explore patients' perceptions of the surgical pathway. This will be analysed from interview transcripts through qualitative analysis using thematic content analysis.
Change in Well Being - Self-efficacy (General Self Efficacy Scale) | Baseline, one week after completion of neo adjuvant treatment, one week before surgery, six weeks after surgery, twelve weeks after surgery
  Self reported measure of Self-efficacy (General Self Efficacy Scale). 10 item questionnaire.Scored 1-4. 1 being "not at all true", 4 being "Exactly True". The total score is calculated by finding the sum of the all items. For the GSE, the total score ranges between 10 and 40, with a higher score indicating more self-efficacy.
Change in Well Being - Mastery (Pearlin Mastery Scale). | Baseline, one week after completion of neo adjuvant treatment, one week before surgery, six weeks after surgery, twelve weeks after surgery
  Mastery (Pearlin Mastery Scale). This consists of seven items designed to assess one aspect of psychological coping resources (Mastery). Example items include, "Sometimes I feel that I am being pushed here and there in life" (reverse-scored) and "What happens to me in the future mostly depends on me." Response options range from 1, strongly disagree, to 7, strongly agree. Score range from 7-28. Higher scores indicate greater mastery.
Fear of Surgery Questionnaire | One week before surgery
  The fear of surgery questionnaire is a valid and reliable eight-item index of surgical fear consisting of two subscales: fear of the short-term consequences of surgery and fear of the long-term consequences. Scoring range 0-100 with 0 being not afraid at all and 100 indicating very afraid.
Post Operative Morbidity - Post Operative Morbidity Score (POMS) | Day 15 post surgery
  Post-operative Morbidity Outcomes: Assessed using the Post-operative Morbidity Score (POMS) at day 15. The POMS is an 18-item tool that addresses morbidity relevant to the post-surgical patient. The subcategories are Pulmonary, Infectious, Renal, Gastrointestinal, Cardiovascular, Neurological, Hematological, Wound and Pain. It is implemented as the morbidity either being present or absent.
Post Operative Morbidity - Post Operative Morbidity Score (POMS) | Day 30 post surgery
  Post-operative Morbidity Outcomes: Assessed using the Post-operative Morbidity Score (POMS) at day 15. The POMS is an 18-item tool that addresses morbidity relevant to the post-surgical patient. The subcategories are Pulmonary, Infectious, Renal, Gastrointestinal, Cardiovascular, Neurological, Hematological, Wound and Pain. It is implemented as the morbidity either being present or absent.
Post Operative Morbidity -Clavien-Dindo Classification of Surgical Outcomes | Day 15 post surgery
  The Clavien-Dindo classification of surgical complications, this consists of 5 grades that rank a post operative complication. grade one being any deviation form the usual post operative course and grade 5 being death.
Post Operative Morbidity -Clavien-Dindo Classification of Surgical Outcomes | Day 30 post surgery
  The Clavien-Dindo classification of surgical complications, this consists of 5 grades that rank a post operative complication. grade one being any deviation form the usual post operative course and grade 5 being death.
Change in Nutritional Status -Assessed using Glasgow Prognostic Score | Baseline, one week after completion of neo adjuvant treatment, one week before surgery,15 days after surgery, 30 days after surgery, six weeks after surgery, twelve weeks after surgery
  The Glasgow Prognostic Score Provides cancer prognosis based on serum biomarkers CRP and Albumin. It is calculated as follows: a score of 0 for normal C reactive protein and albumin levels, score 1 for either an abnormal C reactive protein or abnormal albumin level and score 2 for both abnormal C reactive protein and abnormal albumin levels.
Change in Nutritional Status -Assessed using Foodbook 24 | Baseline, one week after completion of neo adjuvant treatment, one week before surgery, 15 days after surgery, 30 days after surgery, weeks after surgery, twelve weeks after surgery
  Foodbook24 is a Web-based, dietary tool consisting of a 24- hour dietary recall and food frequency questionnaire alongside supplementary questionnaires.
Change in concentration of blood markers of Inflammation- C-Reactive Protein | Baseline, one week after completion of neo adjuvant treatment, one week before surgery, 15 days after surgery, 30 days after surgery, six weeks after surgery, twelve weeks after surgery
  C-Reactive Protein will be assessed at each time point. A level greater that 15mmol/L
Change in concentration of blood markers of Inflammation- White Cell Differential | Baseline, one week after completion of neo adjuvant treatment, one week before surgery, 15 days after surgery, 30 days after surgery, six weeks after surgery, twelve weeks after surgery
  White Cell Differential will be assessed at each time point. Normal range 3.5-10.5 x 109/L

CONTACTS AND LOCATIONS:
Overall Officials: William Robb, MB,BCh,BAO,BA,FRCSI,MD, Principal Investigator — Beaumont Hospital Dublin; Noel McCaffrey, MB,BCh,BAO,BSc,MSc, Study Chair — Dublin City University; Thomas Murphy, MB,BCh,BAO,FRCSI, Study Chair — Mercy University Hospital, Cork; Jarlath Bolger, MB,BCh,BAO,MD, Study Chair — Beaumont Hospital; Pamela Gallagher, Professor of Psychology, Study Chair — Dublin City University; Claire Timon, BSc,PhD, Study Chair — University College Dublin; Jan Sorensen, MSc, MA, Study Chair — Royal College of Surgeons, Ireland
Locations (1):
- Beaumont Hospital, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Loughney L, Bolger J, Tully R, Sorensen J, Bambrick M, Carroll PA, Arumugasamy M, Murphy TJ, McCaffrey N, Robb WB; PERIOP-OG Working Group. The effect of a pre-operative and post-operative exercise programme versus standard care on physical fitness of patients with oesophageal and gastric cancer undergoing neoadjuvant treatment prior to surgery (the PERIOP-OG trial): a randomized controlled trial. Int J Surg. 2024 Oct 1;110(10):6632-6646. doi: 10.1097/JS9.0000000000001663. PMID 38935085
- [Derived] Tully R, Loughney L, Bolger J, Sorensen J, McAnena O, Collins CG, Carroll PA, Arumugasamy M, Murphy TJ, Robb WB; PERIOP OG Working Group. The effect of a pre- and post-operative exercise programme versus standard care on physical fitness of patients with oesophageal and gastric cancer undergoing neoadjuvant treatment prior to surgery (The PERIOP-OG Trial): Study protocol for a randomised controlled trial. Trials. 2020 Jul 13;21(1):638. doi: 10.1186/s13063-020-04311-4. PMID 32660526